CLINICAL TRIAL: NCT03138967
Title: A Phase IV Investigation of Sugammadex in Outpatient Urological Procedures
Brief Title: Investigation of Sugammadex in Outpatient Urological Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-1007
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Malignant Neoplasms of Urinary Tract; Bladder Cancer
Keywords: Malignant neoplasms of urinary tract; Bladder cancer; Outpatient bladder procedures; Outpatient cystoscopy procedure; Transurethral resection of the bladder; TURB; Rocuronium; Rocuronium Bromide; Zemuron; Sugammadex; Neostigmine; Glycopyrrolate
MeSH Terms: conditions — Urologic Neoplasms; Urinary Bladder Neoplasms | interventions — Rocuronium; Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Experimental): Participants to have cystoscopy with bladder tumor resection.
  Rocuronium used to induce the neuromuscular blockade and given in a rapid sequence for endotracheal intubation at a dose of 0.45 mg/kg of Ideal Body Weight. If maintenance is needed for continued relaxation then a dose of 0.15 mg/kg of Ideal Body Weight repeated as necessary.
  Sugammadex administered as a single bolus, intravenous injection. The amount used is based on the patient's weight. A dose of 4 mg/kg used if recovery has reached at least 1-2 post-tetanic counts (PTC) following Rocuronium induced blockade.
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Standard of Care - Neostigmine/Glycopyrrolate (Active Comparator): Participants to have cystoscopy with bladder tumor resection.
  Rocuronium used to induce the neuromuscular blockade and given in a rapid sequence for endotracheal intubation at a dose of 0.45 mg/kg of Ideal Body Weight. If maintenance is needed for continued relaxation then a dose of 0.15 mg/kg of Ideal Body Weight repeated as necessary.
  Neostigmine/Glycopyrrolate administered as a single bolus, intravenous injection. The amount used is based on the patient's weight. Once T1 is at 10% or greater, a dose of 70 mcg/kg of Neostigmine with 14 mcg/kg Glycopyrrolate administered simultaneously over a period of one minute up to 5 mg.
  Interventions: Drug: Rocuronium; Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Rocuronium — Experimental: Sugammadex Participants to have cystoscopy with bladder tumor resection. Rocuronium used to induce the neuromuscular blockade and given in a rapid sequence for endotracheal intubation at a dose of 0.45 mg/kg of Ideal Body Weight. If maintenance is needed for continued relaxation then a dose of 0.15 mg/kg of Ideal Body Weight repeated as necessary.
  Other Names: Rocuronium Bromide; Zemuron
Drug: Sugammadex — Sugammadex administered as a single bolus, intravenous injection. The amount used is based on the patient's weight. A dose of 4 mg/kg used if recovery has reached at least 1-2 post-tetanic counts (PTC) following Rocuronium induced blockade.
  Arms: Sugammadex
Drug: Neostigmine — 70 mcg/kg by vein to reverse the muscle relaxation.
  Arms: Standard of Care - Neostigmine/Glycopyrrolate
Drug: Glycopyrrolate — 14 mcg/kg by vein to reverse the muscle relaxation.
  Arms: Standard of Care - Neostigmine/Glycopyrrolate

SUMMARY:
The goal of this clinical research study is to determine whether using sugammadex, given with a standard muscle relaxation drug during bladder surgeries, improves anesthesia conditions and recovery time.

During some bladder operations, your muscles must be completely relaxed. Muscle relaxation drugs cause the muscles to relax, including the respiratory muscles, and as a result artificial ventilation is needed to help you breathe. Sugammadex and other standard drugs reverse the effect of the muscle relaxation drugs, allowing you to breathe on your own after the operation.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group:

* If you are in Group 1, you will receive sugammadex to reverse the muscle relaxation.
* If you are in Group 2, you will receive the standard of care (neostigmine/glycopyrrolate) to reverse the muscle relaxation.

You and the surgeon will not know which group you have been assigned to. However, the anesthesiologist and study staff will know.

Length of Study:

You will be on study for up to 1 week after the cystoscopy. If you are unable to have the procedure performed, you may be taken off study early.

This is an investigational study. Sugammadex and neostigmine/glycopyrrolate are all FDA approved and commercially available to reverse muscle relaxation. The comparison of these drugs is investigational.

Up to 50 participants will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Procedures:

Before the cystoscopy, we will collect your basic information and medical history. We will take your vital signs and the anesthesiologist will perform routine assessments. This will take about 30-60 minutes to complete.

Before the cystoscopy, you will be given rocuronium to relax your muscles. After the procedure, you will receive either sugammadex or the standard of care to reverse the relaxation.

After you are extubated (the tube is removed from your throat), we will assess how fast the relaxation drugs the anesthesiologist gave you wear off (stop working), using a small monitoring device that will be attached to your wrist. This is the only research test that will be done right after surgery.

If you are still in the hospital 1 day after the cystoscopy, a member of the staff will ask you the series of questions. If you have been sent home, you will be called and you will complete them by phone.

Researchers will also collect information about your cystoscopy procedure and recovery from your medical record. This collection will continue for up to 1 week after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Is scheduled to undergo cystoscopy with bladder resection procedure under general anesthesia requiring neuromuscular relaxation using rocuronium bromide to secure airway and requiring neuromuscular reversal at The University of Texas MD Anderson Cancer Center - Mays Clinic (ACB-outpatient)
2. Male or Females who are >= 18 years of age
3. Classified by the American Society of Anesthesiologists (ASA) as Class I - IV
4. Candidate for use of laryngeal mask airway (LMA)
5. Able to give consent

Exclusion Criteria:

1. Severe renal impairment as measured eGFR less than 30 per institutional laboratory.
2. Females who are pregnant or might be pregnant or are breast-feeding.
3. Females who have been diagnosed with breast cancer and currently taking Toremifene
4. Is known or suspected to have significant hepatic dysfunction, with AST & ALT 3 times above UNL per institutional laboratory.
5. Is known or suspected to have a (family) history of malignant hyperthermia
6. Is known or suspected to have an allergy to opioids, muscle relaxants or other medications used during general anesthesia
7. Is known or suspected to have neuromuscular disorders (ex: myasthenia gravis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Goravanchi, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened within days of their scheduled eligible procedure. Enrolled 50 patients, 4 withdrew, we requested IRB approval to enroll 4 more to maintain statistical power. A total of 54 patients were enrolled in the study, but only 50 were assessed for the primary outcome, 1 participant died before POD-7 follow-up.
Groups:
- Suggamadex or Treatment Group: Sugammadex will be administered as a single bolus, intravenous injection. The amount used is based on the patient's weight. A dose of 4 mg/kg will be used if recovery has reached at least 1-2 post-tetanic counts (PTC) following Rocuronium induced blockade.
- Neostigime/Glycopyrrolate or Standard of Care Group: Neostigmine/Glycopyrrolate will be administered as a single bolus, intravenous injection. The amount used is based on the patient's weight. Once T1 is at 10% or greater, a dose of 70mcg/kg of neostigmine with 14 mcg/kg glycopyrrolate will be administered simultaneously over a period of one minute up to 5 mg.
Period: Overall Study
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group
Started | 26 | 28
Post-operative Day(POD) 1 Follow-up | 25 | 25
Post-operative Day(POD) 7 Follow-up | 25 | 24
Completed | 25 | 24
Not Completed | 1 | 4
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1923 (8.04) | 71.6071 (8.7235) | 69.48 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 18 | 25 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 21 | 43
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 54
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.9385 (5.7725) | 28.7214 (4.766) | 28.34 (5.24)

OUTCOME MEASURES:

1. Primary Outcome: Muscle Recovery Time
Description: The primary outcome is to determine if Sugammadex can improve muscle recovery time, measured by time from administration of neuromuscular blockade reversal to train-of-four ratio of 0.9 in outpatient bladder procedures. It was assessed in the intraoperative period measuring the time from administration of reversal agent to TOF of 0.9 in minutes.
Time Frame: Intraoperatively, up to 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group
Number analyzed (Participants) | 25 | 25
minutes | 2 (0.6455) | 9.24 (7.8755)

2. Secondary Outcome: PostOperative Complications
Description: To determine if Sugammadex can improve post-operative complications for outpatient bladder procedures such as bladder perforation, nausea, vomiting, post-operative intubation and hospital admittance secondary to respiratory complications which was assessed uring follow ups on post-operative day 1 (POD1) and post-operative day 7 (POD7) looking for immediate postoperative complications such as bladder perforation, nausea, vomiting, postoperative intubation and hospital admittance secondary to respiratory complications and readmission within a week post-procedure for any other cause.
Time Frame: Post-operatively, up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group
Number analyzed (Participants) | 25 | 25
Participants | 5 | 7

3. Secondary Outcome: Overall Recovery Time
Description: To determine if Sugammadex can improve overall recovery time, measured by time from end of surgery to the time patient met Discharge Criteria.
Time Frame: Up to 3 hours after end of surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group
Number analyzed (Participants) | 25 | 25
hours | 2.0847 (0.8742) | 2.4727 (2.0447)

ADVERSE EVENTS:
Time Frame: 7 days post surgery
Arm/Group | Suggamadex or Treatment Group | Neostigime/Glycopyrrolate or Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 5/25 | 6/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suggamadex or Treatment Group (N=25) | Neostigime/Glycopyrrolate or Standard of Care Group (N=25)
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suggamadex or Treatment Group (N=25) | Neostigime/Glycopyrrolate or Standard of Care Group (N=25)
Hematuria (Renal and urinary disorders) | 1 | 2
Uncontrolled Hypertension (Cardiac disorders) | 0 | 1
Laceration of penis' skin (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Hematuria with Clot retention (Renal and urinary disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
IV infiltration (Skin and subcutaneous tissue disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03138967/Prot_SAP_000.pdf